CLINICAL TRIAL: NCT07200219
Title: A Quasi-Experimental Study on the Effect of Psychological Performance Strategies Training on Achievement Motivation in Athletes
Brief Title: Psychological Performance Strategies Training to Improve Achievement Motivation in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ladislav Batalik (Other)
Responsible Party: Sponsor-Investigator, Ladislav Batalik, Associate Professor, Department of Physiotherapy and Rehabilitation, Faculty of Medicine, Masaryk University; Department of Rehabilitation, University Hospital Brno, Brno University Hospital
Organization: Brno University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPS-ATH-2025
Record Dates: First submitted 2025-09-26; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Achievement; Athlete; Athletic Performance; Sports

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological Performance Strategies Training (Experimental): Licensed athletes received a structured, supervised psychological performance strategies training program over 4 weeks. The program consisted of 8 modules (two 60-minute sessions per week) covering goal setting, self-talk, emotional control, imagery, automaticity, action orientation, attention control/negative thinking management, and relaxation techniques. Training was delivered in a group setting by qualified instructors.
  Interventions: Behavioral: Psychological Performance Strategies Training
- No Intervention (No Intervention): Licensed athletes assigned to the control group did not receive any psychological training during the 4-week period. They continued their usual academic and training routines without additional intervention.

INTERVENTIONS:
Behavioral: Psychological Performance Strategies Training — A structured 4-week program of psychological performance strategies training delivered to licensed athletes. The program consisted of 8 sessions (twice per week, 60 minutes each) including modules on goal setting, self-talk, emotional control, imagery, automaticity, action orientation, attention control/negative thinking management, and relaxation techniques. Training was conducted in a supervised group format by qualified instructors.
  Arms: Psychological Performance Strategies Training

SUMMARY:
This quasi-experimental study was designed to evaluate whether a structured, four-week psychological performance strategies training program could improve achievement motivation among licensed athletes. Fifty athletes were assigned to an experimental group (n=25) and a control group (n=25). The experimental group received training twice weekly for four weeks, including goal setting, self-talk, emotional control, imagery, automaticity, action orientation, attention control, and relaxation. Achievement motivation was measured at baseline and after the intervention using the Sport-Specific Achievement Motivation Scale.

DETAILED DESCRIPTION:
Achievement motivation is a key determinant of athletic performance, yet few studies have systematically investigated structured psychological skills training in this area. This study aimed to examine the effect of a multi-component psychological performance strategies program on achievement motivation in athletes.

A total of 50 licensed athletes from the Faculty of Sports Sciences, Aksaray University, voluntarily participated. Participants were divided into an experimental group (n=25) and a control group (n=25). The experimental group received supervised psychological performance strategies training, consisting of eight modules delivered over four weeks (two sessions per week, 60 minutes each). Training content included:

* Goal setting
* Self-talk
* Emotional control
* Imagery
* Automaticity
* Taking action
* Attention control and negative thinking management
* Relaxation techniques

The control group did not receive any intervention. Outcome assessment was performed using the Sport-Specific Achievement Motivation Scale, administered at baseline and after the 4-week program.

ELIGIBILITY:
Inclusion Criteria:

* Licensed athletes enrolled at the Faculty of Sports Sciences, Aksaray University
* Age ≥18 years
* Voluntary agreement to participate and provide informed consent
* No prior participation in psychological performance strategy training

Exclusion Criteria:

* Previous exposure to structured sports psychology or psychological skills training programs
* Presence of acute injury, illness, or medical condition preventing participation
* Refusal or inability to provide informed consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Sport-Specific Achievement Motivation total score | Baseline (Week 0) to Post-intervention (Week 4)
  Mean change in the Sport-Specific Achievement Motivation Scale (40 items, 5-point Likert; minimum = 1, maximum = 5; higher scores indicate greater achievement motivation) from baseline to post-intervention. Scores assessed in both arms; between-group comparison based on change scores.

SECONDARY OUTCOMES:
Percent change in Sport-Specific Achievement Motivation total score | Baseline (Week 0) to Post-intervention (Week 4)
  Percent change = [(Post-test - Pre-test) / Pre-test] × 100; calculated using the Sport-Specific Achievement Motivation Scale (40 items, 5-point Likert; minimum = 1, maximum = 5; higher scores indicate greater achievement motivation).
Post-intervention Sport-Specific Achievement Motivation total score | Post-intervention (Week 4)
  Group comparison of Sport-Specific Achievement Motivation Scale total score at Week 4 (40 items, 5-point Likert; minimum = 1, maximum = 5; higher scores indicate greater achievement motivation). Baseline score considered in analysis as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Metin YÜCEANT, PhD, Principal Investigator — Aksaray Üniversitesi Spor Bilimleri Fakültesi, Turkey
Locations (1):
- Aksaray University, Faculty of Sports Sciences, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No